CLINICAL TRIAL: NCT00570310
Title: A Double-Blind, Placebo-Controlled, Enriched-Enrollment, Randomized Withdrawal Study to Evaluate an Optimal Methodology for Conducting Proof of Concept Trials in Patients With Chronic Neuropathic Pain Syndromes Using Pregabalin as a Test Drug
Brief Title: Neuropathic Pain Syndrome Patient Study (MK-0000-072)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-072; 2007_650
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Results first posted 2010-02-05 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-04

CONDITIONS: Neuralgia, Postherpetic; Diabetic Neuropathy; Painful Small-Fiber Neuropathy; Idiopathic Distal Sensory Polyneuropathy
MeSH Terms: conditions — Neuralgia, Postherpetic; Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Active Comparator): Patients in Group A will remain on pregabalin (up to 600 mg/day po) treatment for the entire double-blind period.
  Interventions: Drug: Comparator: pregabalin
- B (Placebo Comparator): Patients in Group B will be treated with placebo.
  Interventions: Drug: Comparator: Placebo (unspecified)

INTERVENTIONS:
Drug: Comparator: pregabalin — pregabalin (up to 600 mg/day by mouth (po)). Duration of Treatment: 6 Weeks
  Arms: A
Drug: Comparator: Placebo (unspecified) — pregabalin Pbo (up to 600 mg/day by mouth (po)). Duration of Treatment: 6 Weeks
  Arms: B

SUMMARY:
The purpose of this study is to determine the best way to conduct clinical trials in patients with neuropathic pain (nerve pain). This study will see if generic pregabalin has any effect on neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient has moderate to severe nerve pain due to one of the following conditions: Postherpetic neuralgia, Painful diabetic neuropathy, Small fiber neuropathy or idiopathic distal sensory polyneuropathy
* Patient is able to complete questionnaires in either English or Spanish
* Patient is at least 18 years of age

Exclusion Criteria:

* Patient is either pregnant or breastfeeding
* Patient has a history of angioedema (swelling beneath the skin surface) or peripheral edema (foot, leg, and/or ankle swelling)
* Patient has a history of congestive heart failure
* Patient has a seizure disorder
* Patient has a history of drug and/or alcohol abuse within the past 1 year
* Patient failed treatment due to lack of pain relief with more than three drugs for nerve pain
* Patient has had cancer (except basal cell carcinoma) within the past two years
* Patient anticipates the need for surgery while participating in the study
* Patient has a reported history of hepatitis B, C, or HIV infection
* Patient has another type of pain that is more painful than the nerve pain
* Patient has generalized anxiety disorder, untreated depression, psychosis, or post-traumatic stress disorder
* Patient is involved in litigation or receives worker's compensation related to nerve pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Hewitt DJ, Ho TW, Galer B, Backonja M, Markovitz P, Gammaitoni A, Michelson D, Bolognese J, Alon A, Rosenberg E, Herman G, Wang H. Impact of responder definition on the enriched enrollment randomized withdrawal trial design for establishing proof of concept in neuropathic pain. Pain. 2011 Mar;152(3):514-521. doi: 10.1016/j.pain.2010.10.050. Epub 2010 Dec 23. PMID 21185118

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Last Patient Entered: 06-Dec-07
  Last Patient Last Visit: 11-Sep-08
  # Sites: 20 sites randomized at least 1 patient.
  21 sites screened at least 1 patient
Pre-assignment Details: All patients were titrated up to the maximum tolerated dose of active treatment (pregabalin) over approximately 12 days. Patient were treated at the maximum tolerated dose until randomization at which time patient were either continued on active treatment or withdrawn from active treatment (i.e. placebo) in a double-blind fashion.
Groups:
- Pregabalin: Patients were treated with pregabalin (up to 600 mg/day by mouth (po)) for the entire double-blind period.
- Placebo: Patients were treated with placebo starting at randomization.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 53 | 51
Completed | 51 | 45
Not Completed | 2 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Pregabalin: Patients who were randomized to pregabalin and were categorized in the primary responder population. Primary responders were defined as having ≥30% decrease in mean of average daily pain intensity during the last 3 days of the pre-randomization maintenance phase relative to baseline.
- Placebo: Patients who were randomized to placebo and were categorized in the primary responder population. Primary responders were defined as having ≥30% decrease in mean of average daily pain intensity during the last 3 days of the pre-randomization maintenance phase relative to baseline.
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.8) | 59.3 (11.0) | 60.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 14 | 22
  Male | 22 | 18 | 40
Body Mass Index [Mean (Full Range); unit: kilograms/meter^2] | 32.6 [20.9 to 49.3] | 31.3 [18.5 to 49.5] | 31.9 [18.5 to 49.5]

OUTCOME MEASURES:

1. Primary Outcome: Daily Evening Patient Reported Pain Intensity Scores
Description: Change from mean of last 3 days of maintenance period to last 3 days of double-blind period; Pain Intensity was rated on a 0-10 numeric rating scale (NRS: 0=no pain, 10=worst pain you can imagine)
Time Frame: Baseline and 6 Weeks
Population: Patients who had a ≥30% decrease in mean of average daily pain intensity during the last 3 days of the maintenance phase relative to baseline.
Measure: Least Squares Mean (Full Range); unit: Units on a Scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 30 | 32
Units on a Scale | 0.14 [-2.00 to 4.33] | 1.57 [-1.83 to 8.00]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.003, ANOVA — 1-sided, alpha = 0.05; Mean Difference (Final Values) = -1.42, 90% CI [-2.25 to -0.60] — Primary Hypothesis: In 'primary responder population', pregabalin is superior to placebo in maintaining pain control measured by change (3-day average: end of the randomization period versus end of maintenance period) in evening pain intensity

2. Secondary Outcome: 'Time to Efficacy Failure' During the Randomized Withdrawal Portion of the Study
Description: Time to treatment failure (3 day mean of average 24 hour pain intensity ≥ 4 with at least a 30% increase relative to the last 3 days prior to randomization)
Time Frame: 6 Weeks
Population: Primary Responders: ≥30% decrease in mean of average daily pain intensity during the last 3 days of the maintenance phase relative to baseline.
Measure: Least Squares Mean (Full Range); unit: Days
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 30 | 32
Days | 15.54 [3 to 21] | 7.87 [3 to 21]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — 1-sided, alpha = 0.05; Mean Difference (Final Values) = 7.67, 95% CI [5.26 to 10.08]

ADVERSE EVENTS:
Time Frame: The reported AEs were collected after patients were randomized to the double-blind withdrawal period of the study. AEs that were collected prior to randomization are not reported in this document.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/53
Other Adverse Events (participants affected / at risk) | 37/51 | 36/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=51) | Placebo (N=53)
Arrhythmia (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=51) | Placebo (N=53)
Vertigo (Ear and labyrinth disorders) | 3 | 0
Blindness (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Eye Irritation (Eye disorders) | 0 | 1
Eye Pain (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 3 | 4
Visual Acuity Reduced (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dry Mouth (Gastrointestinal disorders) | 6 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Energy Increased (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 4
Gait Disturbance (General disorders) | 1 | 1
Oedema Peripheral (General disorders) | 5 | 3
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Gastric Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Localised Infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Joint Sprain (Injury, poisoning and procedural complications) | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0
Blood Glucose Decreased (Investigations) | 0 | 1
Blood Glucose Increased (Investigations) | 1 | 0
Weight Increased (Investigations) | 3 | 2
Fluid Retention (Metabolism and nutrition disorders) | 0 | 1
Increased Appetite (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Ataxia (Nervous system disorders) | 0 | 1
Balance Disorder (Nervous system disorders) | 2 | 1
Cluster Headache (Nervous system disorders) | 1 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 1
Disturbance In Attention (Nervous system disorders) | 2 | 2
Dizziness (Nervous system disorders) | 10 | 11
Drooling (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Hypersomnia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypokinesia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 1
Memory Impairment (Nervous system disorders) | 3 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 1
Peroneal Nerve Palsy (Nervous system disorders) | 1 | 0
Poor Quality Sleep (Nervous system disorders) | 1 | 0
Restless Legs Syndrome (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 0 | 1
Sinus Headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 8 | 7
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 2 | 1
Abnormal Dreams (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Bradyphrenia (Psychiatric disorders) | 0 | 2
Confusional State (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Euphoric Mood (Psychiatric disorders) | 1 | 1
Hallucination (Psychiatric disorders) | 1 | 1
Initial Insomnia (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 2
Libido Decreased (Psychiatric disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 1
Urinary Hesitation (Renal and urinary disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Photodermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Peripheral Coldness (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.